CLINICAL TRIAL: NCT03301350
Title: A Phase II Study of Neoadjuvant Carboplatin/Paclitaxel Followed by Dose-Dense Doxorubicin/Cyclophosphamide in Patients With Hormone Receptor Negative, HER2 Receptor Negative Breast Cancer
Brief Title: Neoadjuvant Carbo/Paclitaxel Followed by Doxorubicin/Cyclophosphamide in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16112; NCI-2017-01705 (Registry Identifier: NCI CTRP); 2017-0547 (Other: UW IRB); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 11/26/2019 (Other: UW Madison)
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Carboplatin; Paclitaxel; Doxorubicin; liposomal doxorubicin; Cyclophosphamide; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant Chemotherapy (Experimental): Regimen A (cycles 1-4):
  Paclitaxel 80 mg/m2; administer intravenously on day 1, 8, 15 of cycles 1, 2, 3, 4 (every 3 weeks) Carboplatin AUC=2 (dose calculation by determining creatine clearance with Cockroft Gault using adjusted body weight); administer intravenously on day 1, 8, 15 of cycles 1, 2, 3, 4 (every 3 weeks)
  Regimen B (cycles 5-8):
  Doxorubicin 60 mg/m2; administer intravenously on day 1 of cycles 5, 6, 7, 8 (every 2 weeks) Cyclophosphamide 600 mg/m2; administer intravenously on day 1 of cycles 5, 6, 7, 8 (every 2 weeks) Pegfilgrastim (for use on Doxorubicin/Cyclophosphamide cycles only), filgrastim, or biosimilar support on day 2 - 3 of cycles 5, 6, 7, 8 (every 2 weeks)
  There is a one week break between the end of cycle 4 and the beginning of cycle 5.
  Regimen C:
  Surgical intervention for management of breast cancer diagnosis; procedure and timing as determined by surgical team.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Pegfilgrastim; Drug: Filgrastim

INTERVENTIONS:
Drug: Carboplatin — Carboplatin is a platinum compound alkylating agent which covalently binds to DNA; interferes with the function of DNA by producing interstrand DNA cross-links.
Drug: Paclitaxel — Paclitaxel promotes microtubule assembly by enhancing the action of tubulin dimers, stabilizing existing microtubules, and inhibiting their disassembly, interfering with the late G2 mitotic phase, and inhibiting cell replication. In addition, the drug can distort mitotic spindles, resulting in the breakage of chromosomes. Paclitaxel may also suppress cell proliferation and modulate immune response.
Drug: Doxorubicin — Inhibition of DNA and RNA synthesis by intercalation between DNA base pairs by inhibition of topoisomerase II and by steric obstruction. Doxorubicin intercalates at points of local uncoiling of the double helix. Although the exact mechanism is unclear, it appears that direct binding to DNA (intercalation) and inhibition of DNA repair (topoisomerase II inhibition) result in blockade of DNA and RNA synthesis and fragmentation of DNA. Doxorubicin is also a powerful iron chelator; the iron-doxorubicin complex can bind DNA and cell membranes and produce free radicals that immediately cleave the DNA and cell membranes.
  Other Names: Adriamycin; Doxil; Caelyx; Myocet
Drug: Cyclophosphamide — Cyclophosphamide is an alkylating agent that prevents cell division by cross-linking DNA strands and decreasing DNA synthesis. It is a cell cycle phase nonspecific agent. Cyclophosphamide also possesses potent immunosuppressive activity. Cyclophosphamide is a prodrug that must be metabolized to active metabolites in the liver.
  Other Names: cytophosphane
Drug: Pegfilgrastim — Pegfilgrastim provides growth factor support in a single dose. It stimulates bone marrow to create neutrophils for patients undergoing chemotherapy.
Drug: Filgrastim — Filgrastim provides growth factor support in multiple doses. It stimulates bone marrow to create neutrophils for patients undergoing chemotherapy.

SUMMARY:
This is a phase II single-arm, open-label, prospective study to evaluate the efficacy of the low dose weekly Carboplatin/Paclitaxel followed by dose-dense Doxorubicin/Cyclophosphamide in subjects with triple-negative breast cancer in neoadjuvant settings.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed invasive breast cancer which meets the following criteria:

   1. Estrogen Receptor (ER) and Progesterone Receptor (PR)-negative as defined by local standard clinical immunohistochemistry (IHC) < 1%.
   2. HER2-negative using local standard testing. Negative is defined as IHC 0 or 1+ (if 2+, must reflex to ISH method). If ISH method is used, ratio < 2 is considered negative.
   3. Clinical tumor size of at least 2.1 cm (T2) by palpation or imaging, regardless of the ipsilateral regional lymph node status, or any tumor size but with ipsilateral regional lymph nodes involved by the tumor (any T if ipsilateral regional node positive). Subjects with inflammatory breast cancer are eligible. If bilateral breast cancer is present, the subject is eligible if the contralateral tumor is DCIS only (without any invasive disease on biopsy) or another invasive breast cancer of any size that is also ER, PR and HER2 negative.
   4. Any radiographic abnormal ipsilateral regional lymph nodes or any clinically concerning ipsilateral regional lymph nodes with the exception of internal mammary nodes should be sampled with percutaneous biopsy, but no sentinel axillary lymph node mapping/biopsy is allowed before chemotherapy. If clinically node negative (cNO), pre-chemotherapy ipsilateral sentinel axillary lymph node mapping/biopsy is not allowed.
2. Candidate for neoadjuvant chemotherapy.
3. Age > 18 years and < 75 years
4. ECOG Performance Status < 1.
5. Left ventricular ejection fraction (LVEF) ≥ LLN (per institutional normal) determined by
6. Adequate organ and marrow function as determined by study protocol
7. Non Pregnant. Women of childbearing potential must have a negative pregnancy test (HCG serum or urine) within 30 days prior to study registration and to be repeated if not done within 7 days of starting chemotherapy.

   1. Female subjects must meet one of the following:

      * Natural postmenopausal before the screening visit defined as no menses at any time in the preceding 12 consecutive months, or
      * Prior bilateral oophorectomy or bilateral tubal ligation, or
      * If they are of childbearing potential, agree to practice two effective methods of contraception per discussion with the treating physicians from
   2. Male subjects, even if surgically sterilized (i.e., status post vasectomy) must agree to one of the following:

      * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose, or
      * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
8. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Prior chemotherapy or radiation therapy for invasive breast cancer within 6 months before registration.
2. Prior investigational drugs or interventions for invasive breast cancer within 6 months before registration are not allowed. Prior participation in window-of-opportunity trials without therapeutic intent is allowed if intervention is no more than 3 weeks duration.
3. Stage IV metastatic breast cancer
4. History of allergic reactions attributed to compounds of similar chemical composition to chemotherapy to be used in this study.
5. Breastfeeding women. Cytotoxic chemotherapy is drug with the potential for teratogenic or abortifacient effects. Due to unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cytotoxic chemotherapy, breastfeeding should be discontinued.
6. Baseline peripheral neuropathy of severity > grade 1
7. Other invasive cancer diagnosis within the past 5 years other than non-melanoma skin cancer.
8. Prior axillary lymph node dissection that preclude patient from surgical evaluation of axillary lymph node status.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Wisinski, MD, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - Swedish American Hospital, Rockford, Illinois
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Columbia St. Mary's Cancer Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center Wausau, Wausau, Wisconsin

REFERENCES:
- See also: UW Carbone Cancer Center home page — http://www.uwhealth.org/uw-carbone-cancer-center/47424

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 participants were assigned, but only 28 participants started treatment
Groups:
- Neoadjuvant Chemotherapy: Participants receive Paclitaxel and Carboplatin AUC=2 on days 1, 8, 15 of cycles 1, 2, 3, 4 (every 3 weeks).
  There is a one week break between the end of cycle 4 and the beginning of cycle 5.
  Participants receive Doxorubicin and Cyclophosphamide on day 1 of cycles 5, 6, 7, 8 (every 2 weeks). Participants also receive Pegfilgrastim, filgrastim, or biosimilar support on day 2 - 3 of cycles 5, 6, 7, 8 (every 2 weeks)
  Participants undergo surgical intervention for management of breast cancer diagnosis; procedure and timing as determined by surgical team.
Period: Overall Study
Arm/Group | Neoadjuvant Chemotherapy
Started | 29
Completed | 21
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Pt withdrawn per DSMC request | 1
Not completed — completed all chemo cycles, however died prior to definitive surgery | 1
Not completed — no detail provided | 1

BASELINE CHARACTERISTICS:
Population: 1 participant withdrew after being assigned but prior to treatment. Characteristics were collected for baseline hence 29 baseline participants being reported
Groups:
- Neoadjuvant Chemotherapy: Paclitaxel (cycles 1-4):
  Doxorubicin, Cyclophosphamide, and Pegfilgrastim (cycles 5-8):
  Surgical intervention for management of breast cancer diagnosis; procedure and timing as determined by surgical team.
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 29
Age, Customized [Count of Participants; unit: Participants]
  30-39 | 5
  40-49 | 7
  50-59 | 12
  60-69 | 3
  70-79 | 1
  80-89 | 1
  Unknown | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Pathologic Complete Response (pCR) Rate
Description: pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy. pCR will be assessed according to RECIST 1.1 criteria. The point estimate of the primary efficacy endpoint pCR and its exact 95% confidence intervals (CI) will be calculated. In evaluating pCR, subjects with missing data will be considered non-responders.
Time Frame: Up to 2 years
Population: 4 participants did not reach the timepoint at which pCR was measured, therefore are not counted in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 24
Participants | 8

2. Secondary Outcome: Number of Cycles of Chemotherapy Administered
Description: To evaluate the number of cycles low dose weekly Carboplatin/Paclitaxel regimen administered. Simple descriptive statistics will be used to describe the number of cycles of chemotherapy administered.
Time Frame: Week 12 to week 18 to account for possible delays
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 28
Participants
  4 complete cycles | 25
  Less than 1 cycle | 3

3. Secondary Outcome: Total Dose of Chemotherapy Administered
Description: To evaluate the total dose of weekly Carboplatin/Paclitaxel regimen administered. Simple descriptive statistics will be used to describe the dose amount of chemotherapy administered.
Time Frame: Week 12 to week 18 to account for possible delays
Population: 2 participants were withdrawn from study prior to completing carbo-paclitaxel; thus, have not been included in this measure
Measure: Number; unit: doses administered
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 26
doses administered
  Carboplatin dose AUC of 2.0 - full dose | 285
  paclitaxel dose: 80 mg/m2 - full dose | 279
  Carboplatin reduced dose AUC 1.6 | 15
  Carboplatin reduced dose AUC 1.5 | 2
  Paclitaxel - reduced dose | 23

4. Secondary Outcome: Delays of Administered Chemotherapy
Description: To evaluate the delays of low dose weekly Carboplatin/Paclitaxel regimen administered. Simple descriptive statistics will be used to describe the delays of chemotherapy administered.
Time Frame: Week 12 to week 18 to account for possible delays
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 26
Participants
  Participants with no delays | 12
  Participants with single 1 week delay | 7
  Participants with single 2 week delay | 3
  Participants with more than 1 delay | 4

5. Secondary Outcome: Number of Treatment-related Toxicities Experienced by Participants
Description: Count of any treatment-related toxicities from the low dose weekly Carboplatin/Paclitaxel regimen. Will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to week 12
Measure: Number; unit: treatment related toxicities
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 28
treatment related toxicities
  Neutrophil count decreased | 26
  Anemia | 27
  Platelet count decreased | 22
  White blood cells decreased | 25
  ALT increased | 9
  AST increased | 8
  Creatinine increased | 2
  Bilirubin increased | 1

6. Secondary Outcome: Recurrence-free Survival (RFS)
Description: To evaluate two-year RFS after treatment with this neoadjuvant regimen. Count of participants without evidence for local-regional or distant relapse, second primary, or death will be reported.
Time Frame: Up to 2 years
Population: 4 participants did not reach the timepoint at which RFS was measured, therefore are not counted in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 24
Participants
  No evidence of disease | 18
  Alive, recurrent disease | 2
  Deceased, recurrent disease | 2
  Alive, unknown disease status | 2

7. Secondary Outcome: Overall Survival (OS)
Description: To evaluate the two-year overall survival after treatment with this neoadjuvant regimen. Count of participants who achieved 2 year OS is reported.
Time Frame: Up to 2 years
Population: 3 participants did not reach the timepoint at which OS was measured, therefore are not counted in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemotherapy
Number analyzed (Participants) | 25
Participants
  2 year survival | 22
  Deceased | 3

ADVERSE EVENTS:
Time Frame: 2 years from starting study treatment
Description: Other (Not Including Serious) Adverse Events were not collected/monitored at collaborating site for 18 of the participants; therefore, there is no data to report and the number assessed is most accurately represented as 10 at risk for Other Adverse Events.
Arm/Group | Neoadjuvant Chemotherapy
All-Cause Mortality (participants affected / at risk) | 3/28
Serious Adverse Events (participants affected / at risk) | 17/28
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemotherapy (N=28)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Atrial fibrilation (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Abdomincal pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 15 (15)
platelet count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemotherapy (N=10)
Anemia (Blood and lymphatic system disorders) | 10 (39)
Neutrophil count decreased (Investigations) | 10 (33)
Platelet count decreased (Investigations) | 8 (18)
White blood cell decreased (Investigations) | 10 (53)
Nausea (Gastrointestinal disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 8 (8)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (7)
Alanine aminotransferase increased (Investigations) | 5 (5)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 9 (9)
Creatinine increased (Investigations) | 2 (3)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Fatigue (General disorders) | 10 (11)
Fever (General disorders) | 5 (5)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Localized edema (General disorders) | 3 (3)
Edema face (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 5 (5)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Nail discoloration (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Dry eye (Eye disorders) | 2 (2)
Conjuntivitis infective (Eye disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 3 (3)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Bilirubin increased (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Complete AE data was not collected; approximately 40% of participants are represented in the data reported in the Adverse Events section. Some enrolling sites have been chronically under- and un-staffed for 2+ years, and have not been able to address the coordinating center's numerous queries related to AE data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT03301350/Prot_SAP_000.pdf